CLINICAL TRIAL: NCT05615116
Title: Clinical Study on the Distribution of Digestive Tract Microbiota Before and After Ileocecal Resection in Crohn's Disease
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shanghai 10th People's Hospital (Other)
Responsible Party: Principal Investigator, Huanlong Qin, Professor, Shanghai 10th People's Hospital
Other Study IDs: xkkb-2022
Record Dates: First submitted 2022-11-05; First posted 2022-11-14 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Crohn Disease; Microtia; Ileocecal; Lesion
MeSH Terms: conditions — Crohn Disease; Congenital Microtia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Before ileocecal resection: Patients diagnosed with Crohn's disease after comprehensive evaluation of clinical symptoms, endoscopic features, radiological manifestations and histological features were recruited，and the patients were admitted for right hemicolectomy
- After ileocecal resection: Patients diagnosed with Crohn's disease after comprehensive evaluation of clinical symptoms, endoscopic features, radiological manifestations and histological features were recruited，and the patients underwent reversal of ileostoma after right hemicolectomy

SUMMARY:
In this study, the microbiota sequencing was used to investigate the changes of microbiota in the terminal ileum and the middle part of ascending colon, the mesenteric adipose tissue of ileum and ascending mesocolon, and oral cavity of patients with Crohn's disease before and after ileocecal resection, so as to further explore the role of ileocecal region in inducing remission of disease.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of Crohn's disease

Exclusion Criteria:

Serious oral diseases (e.g. dental caries, periodontal disease) Other acute or chronic gastrointestinal diseases Probiotics or prebiotic consumption and antibiotic use within 1 month

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Crohn's patients before and after ileocecal resection were divided into two groups， the information of these individuals will be analyzed and some conclusions will be drawn.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-11-15 (Estimated); Primary Completion 2023-03-15 (Estimated); Study Completion 2023-03-15 (Estimated)

PRIMARY OUTCOMES:
Microbial changes of intestinal mucosa | 6 month
  Explore the microbial changes in the mucosa of the terminal ileum and the middle segment of the ascending colon in patients with Crohn's disease before and after ileocecal resection through metagenomic analysis

SECONDARY OUTCOMES:
Microbial changes of mesenteric adipose tissue | 6 month
  Explore the microbial changes in the mesenteric adipose tissue of the terminal ileum and the middle segment of the ascending colon in patients with Crohn's disease before and after ileocecal resection through metagenomic analysis

OTHER OUTCOMES:
Microbial changes of oral cavity | 6 month
  Explore the microbial changes in the buccal region of oral cavity in patients with Crohn's disease before and after ileocecal resection through metagenomic analysis

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai 10th People's Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided